CLINICAL TRIAL: NCT07102199
Title: Effectiveness of Differently Sequenced Attentional Focus Instructions in a Home Exercise Program for Non-Specific Neck Pain: A Randomized Controlled Single-Blind Trial
Brief Title: Effect of Attentional Focus Order in Home Exercise for Neck Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Büşra Tamgüç (Other)
Collaborators: Istanbul Nisantasi University (Other)
Responsible Party: Sponsor-Investigator, Büşra Tamgüç, Physiotherapist, Research Assistant, Bahçeşehir University
Organization: Bahçeşehir University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SBETKK2025-4
Record Dates: First submitted 2025-07-21; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Neck Pain; Motor Learning; Home Exercise Program
Keywords: attentional focus; mechanical neck pain; craniovertebral angle
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: This study has a randomized, controlled, single-blind, prospective study design.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IFO-First (Experimental): Participants included in the study will follow a home exercise program for 3 days a week for 4 weeks, in accordance with the instructions given to their groups. The IFO-First group will first receive internal attention focus instructions, then external attention focus.
  Interventions: Other: Internal focus of attention instructions- First; Other: Home exercises
- EFA-Firts (Experimental): Participants included in the study will follow a home exercise program for 3 days a week for 4 weeks, in accordance with the instructions given to their groups. The EFO-First group will first receive external focus instructions, then internal focus of attention instructions.
  Interventions: Other: External focus of attention instructions- First; Other: Home exercises
- CG (Active Comparator): Participants included in the study will follow a home exercise program without any instructions, 3 days a week for 4 weeks.
  Interventions: Other: Home exercises

INTERVENTIONS:
Other: Internal focus of attention instructions- First — Participants first received internal focus instructions, directing their attention to their own body, followed by external focus instructions.
  Arms: IFO-First
Other: External focus of attention instructions- First — Participants first received internal focus instructions, directing their attention to their own body, followed by external focus instructions.
  Arms: EFA-Firts
Other: Home exercises — Participants' home exercise program includes cervical and scapulothoracic stabilization exercises and self-mobilization exercises with the self-sustained natural apophyseal glide (SNAG) method.

SUMMARY:
According to the International Association for the Study of Pain's 2017 terminology, neck pain is described as an unpleasant sensory and emotional experience originating in the cervical region and potentially radiating toward the scapular area, typically linked to actual or potential tissue injury. Although research on how attentional focus instructions influence postural control remains limited, existing findings suggest that the sequence in which these instructions are delivered can impact sensory processing during postural control assessments. These observations raise compelling questions about the potential benefits of using attentional focus strategies in a structured, sequential manner during neck pain treatment. To date, however, no study has investigated how varying the order of attentional focus cues within a home exercise program affects individuals with non-specific neck pain. This study aimed to fill that gap by evaluating the clinical effectiveness of a home-based exercise protocol utilizing attentional focus instructions in different sequences. The primary outcome was disability level, measured by the Neck Disability Index (NDI). Secondary outcomes included pain intensity assessed via the Visual Analog Scale (VAS), craniovertebral angle (CVA) via photogrammetry, pressure pain threshold (PPT), cervical joint range of motion, dizziness-related disability (Dizziness Handicap Inventory), and the endurance of neck flexor and extensor muscles.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 40 years
* A craniovertebral angle of 53 degrees or less
* A Visual Analog Scale score greater than 3 for pain in the neck and shoulder areas
* Experiencing head and neck pain for a duration exceeding three months
* A Neck Disability Index score ranging from 5 to 24
* A positive result on the cervical flexion-rotation test
* A body mass index within the range of 18.5 to 25 kg/m²
* No history of injury to the neck, trunk, or upper and lower extremities in the past six months

Exclusion Criteria:

* A positive result on the Spurling test
* Reduced or absent reflex responses in the upper extremities,
* Referred pain scoring greater than 7 on the Visual Analog Scale in the affected dermatome
* Diagnosis of cervical spinal stenosis
* Diagnosis of an autoimmune disorder
* Previous surgical intervention in the cervical or shoulder region
* A positive result on the Vertebrobasilar insufficiency test
* Presence of any musculoskeletal deformity or abnormality
* Inability to carry out functional activities due to visual, auditory, vestibular, or neurological impairments
* Neck pain associated with malignancy or structural abnormalities
* Clinical presentation consistent with a capsular pattern suggestive of arthritis, or the presence of a severe psychological disorder
* Current pregnancy
* Participation in any form of exercise-based treatment or physiotherapy within the last three months

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index (NDI) | The assessment will be performed at two time points: baseline and 4 weeks after the intervention.
  The Neck Disability Index (NDI) was used to assess disability resulting from neck pain. The NDI consists of 10 items: four addressing subjective symptoms (pain intensity, headache, concentration, and sleeping), and six assessing activities of daily living (personal care, lifting, reading, work activities, driving, and recreation). Each item is scored on a scale from 0 to 5, with total scores ranging from 0 (no disability) to 50 (maximum disability); lower scores indicate less disability. According to the literature, the minimal clinically important difference (MCID) for the NDI has been reported to be 7 points (Abbott, 2014).

SECONDARY OUTCOMES:
Pain Intensity Based on Visual Analog Pain Scale (VAS) | The assessment will be performed at two time points: baseline and 4 weeks after the intervention.
  The Visual Analog Scale (VAS) will be used to assess the intensity of pain experienced by patients with neck pain during movement and at rest. According to the VAS, patients are asked to rate their perceived pain intensity on a scale from 0 to 10, where "0" represents "no pain" and "10" represents "the worst pain imaginable.
Dizzines Handicap Inventory | The assessment will be performed at two time points: baseline and 4 weeks after the intervention.
  The Dizziness Handicap Inventory (DHI) will be used to assess patients' quality of life. This scale consists of 25 items that evaluate the aggravating factors related to dizziness and balance disorders, as well as the emotional and functional consequences of vestibular system diseases. The DHI is a self-reported measure with three subscales: functional, emotional, and physical. Patients rate their perceived dizziness-related disability by responding to each item with "Yes," "Sometimes," or "No." Responses are scored as follows: No = 0, Sometimes = 2, and Yes = 4. The total score ranges from 0 to 100, with higher scores indicating greater perceived disability. Patients who score above 10 are recommended to be referred to balance specialists for further evaluation.
Craniovertebral angle measurement | The assessment will be performed at two time points: baseline and 4 weeks after the intervention.
  The craniovertebral angle is defined as the angle formed at the intersection of a line drawn from the tragus of the ear to the C7 vertebra and a horizontal reference line. This angle is commonly used to assess forward head posture. As the angle increases, the degree of forward inclination of the head over the neck also increases. In this study, craniovertebral angle measurements of the participants will be evaluated using a photogrammetric method. For this measurement, markers will be placed on the C7 vertebra and the tragus of the ear, and images of the participants will be captured from both the frontal and sagittal planes.
Pressure Pain Threshold Measurement (PPT) | The assessment will be performed at two time points: baseline and 4 weeks after the intervention.
  The tip of the algometer will be placed perpendicular to the skin, between the acromion and C7, at the midpoint of the upper trapezius muscle, and pressure will be applied at a rate of 1 kg/cm2/s. After an explanation of the measurement and a demonstration of the thenar region of the hand, 3 consecutive PPT measurements will be made at each position, with a 30-second rest between measurements. The average of the PPT measurements will be recorded and the PPT will be evaluated bilaterally.
Cervical Joint Range of Motion Measurement | The assessment will be performed at two time points: baseline and 4 weeks after the intervention.
  Cervical joint range of motion will be measured using a digital goniometer. The assessment will be conducted with the participant seated comfortably on a chair, with both feet flat on the ground, hips and knees positioned at a 90° angle, and only the heels touching the back of the chair. After setting the goniometer to a neutral position, the participant will be instructed to move their head in a standardized manner as far as possible in each direction: flexion, extension, right lateral flexion, left lateral flexion, right rotation, and left rotation. The measurement results will be recorded.
Endurance Test for Neck Flexors | The assessment will be performed at two time points: baseline and 4 weeks after the intervention.
  For endurance testing of the neck flexors, the patient will be asked to chin-in isometrically and then lift the occiput off the surface of the bed while lying supine, both knees flexed, and feet together. The patient will then be instructed to hold the head in this elevated position for as long as possible without assistance. A stopwatch will be used to record the duration of this isometric neck flexion. This phase will be repeated twice with a five-minute interval between each repetition, and the average of the two measurements will be used for data analysis.
Endurance Test for Neck Extensors | The assessment will be performed at two time points: baseline and 4 weeks after the intervention.
  In the prone position, the patient will be instructed to extend their neck over the edge of the couch while securing their upper torso and cervico-thoracic region to the couch. The patient will then chin-in from this neutral position. A stopwatch will be used to record their times in seconds. This phase will be repeated twice with a five-minute interval between each repetition, and the average of the two measurements will be used for data analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Nişantaşı University, Istanbul, Sarıyer, Turkey (Türkiye)